CLINICAL TRIAL: NCT02110823
Title: Single Ventricle Reconstruction Extension Study (A Study Conducted by the Pediatric Heart Network)
Brief Title: Single Ventricle Reconstruction Extension Study (SVR II) - Pediatric Heart Network
Acronym: SVRII
Status: Active, not recruiting | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: U10HL068270-4a; U10HL068270 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Heart Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The SVR II study will collect biological specimens to bank in an established biorepository as a resource for future, hypothesis-driven studies from families who provide separate informed consent. When possible, blood will be drawn, processed, and stored in such a way as to permit both genetic studies and studies of serum biomarkers. The intent is to obtain blood from study subjects and parents (i.e., "trios"). When obtaining blood is not possible, however, saliva will be obtained so that at least genetic information can be stored for future studies.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Single Ventricle Reconstruction (SVR) Trial looked at how infants with single ventricle heart defects did after the first stage of surgery (Norwood operation). Infants enrolled in the trial got one of two kinds of shunts during the Norwood; a modified Blalock-Taussig shunt (MBTS) or right ventricle to pulmonary artery shunt (RV-to-PA shunt).

The purpose of this study is to learn if children (2-6 years of age) who were enrolled in the SVR Trial do better with one of the two shunts (MBTS or RV-to-PA) in the years after surgery.

DETAILED DESCRIPTION:
Among critical congenital heart lesions, hypoplastic left heart syndrome (HLHS) and related single right ventricle (RV) anomalies are associated with the highest morbidity and mortality. The first stage in palliation for patients with these defects is the Norwood procedure. The essential components of the Norwood procedure include (1) an atrial septectomy, (2) anastomosis of the proximal pulmonary artery to the aorta with homograft augmentation of the aortic arch, and (3) establishment of a source of pulmonary blood flow, with either a modified Blalock-Taussig shunt (MBTS) or the right ventricle to pulmonary artery (RV-to-PA) shunt. In May 2005, the Pediatric Heart Network began a multi-center, randomized trial, the Single Ventricle Reconstruction (SVR) Trial, comparing outcomes in subjects with HLHS or other single RV anomalies palliated using the Norwood procedure with either a MBTS or the RV-to-PA shunt. The primary outcome of this trial was freedom from death or cardiac transplantation by 12 months post-randomization.

The Single Ventricle Reconstruction Extension (SVR II) Study is an extension of the SVR Trial that compares clinical outcomes and RV performance following the RV-to-PA shunt versus MBTS modifications of the Norwood procedure in subjects at 6 years post-randomization. Data is collected annually between ages 2 and 6 years, as well as before and after the Fontan surgery. Vital status and medical history is ascertained annually until the last enrolled subject is 6 years old. Data is obtained through medical record review, phone interview with the parent or guardian, electrocardiography (ECG), core laboratory analysis of echocardiographic images and Holter monitors, and completion of questionnaires regarding neurodevelopmental outcomes, behavior, health-related quality of life, and family functioning. The primary outcome variable in SVR II will be freedom from death or cardiac transplantation at 6 years post-randomization. All subjects who were randomized in the SVR trial will be included in analysis of this endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Randomized subject in the Single Ventricle Reconstruction Trial

Exclusion Criteria:

* No subjects enrolled in the the original SVR Trial will be excluded from analysis of the primary endpoint

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Follow up of subjects originally enrolled in the SVR trial
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from death and cardiac transplantation at 6 years post-randomization. | Assessed annually until the last enrolled subject reaches 6 years of age.

SECONDARY OUTCOMES:
Direct and indirect measures of right ventricle (RV) systolic and diastolic function. | Pre-Fontan, and 6 years of age
  * RV ejection fraction by echocardiogram pre-Fontan and at 6 years.
  * RV fractional area change pre-Fontan and at 6 years post-randomization.
  * Severity of tricuspid regurgitation by echocardiogram pre-Fontan and at 6 years.
  * Heart Failure Class pre-Fontan and at 3, 4, 5, and 6 years.
  * Somatic growth pre-Fontan and annually from ages 2-6 years.
6 years post randomization | post procedure up to 6 years post randomization
Incidence of arrhythmias. | Assessed once, at 6 years of age
  * Diagnosis of ventricular arrhythmias by 6 years.
  * Diagnosis of atrial arrhythmias by 6 years.
Neurodevelopment. | Questionnaires completed at ages 3, 4, 5, and 6 years
  Ages & Stages Questionnaires (ASQ)
Behavior | Questionnaires completed at ages 3, 4, 5, and 6 years
  * Behavior Assessment System for Children, Second Edition (BASC-2)
  * Vineland Adaptive Behavior Scales
Health-related quality of life | Questionaires completed at ages 3, 4, 5 and 6 years
  * Pediatric Quality of Life Inventory (PedsQL)
  * Children's Health Questionnaire Parent Form 50-Item (CHQ-PF50) Physical and Psychosocial Function Summary
Family function | Questionnaires completed at ages 3, 4, 5, and 6 years
  Impact on Family Scale Functional States II-R

REFERENCES:
- [Derived] Dolgner SJ, Tjoeng YL, Chan T. Analysis of the Single Ventricle Reconstruction Trial Using Restricted Mean Survival Time and Shunt Type Received. J Am Heart Assoc. 2022 Sep 20;11(18):e025978. doi: 10.1161/JAHA.122.025978. Epub 2022 Sep 8. No abstract available. PMID 36073629